CLINICAL TRIAL: NCT06257017
Title: Surveillance of the Genetic Signature in Circulating Tumor DNA for Guiding Adjuvant Chemotherapy in Urothelial Carcinoma: A Pilot Randomized Controlled Trial
Brief Title: Surveillance of the Genetic Signature in Circulating Tumor DNA for Guiding Adjuvant Chemotherapy in Urothelial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yung NA (Other)
Collaborators: Pamela Youde Nethersole Eastern Hospital (Other); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Yung NA, Clinical Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HKURO202401
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Muscle-Invasive Bladder Carcinoma
Keywords: circulating tumor DNA; ctDNA; molecular residual disease
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine plus cisplatin chemotherapy arm (GC arm) (Experimental): Patients in this group will receive adjuvant chemotherapy of gemcitabine and cisplatin, prior to radiological progression
  Interventions: Drug: gemcitabine; Drug: Cisplatin
- Standard management arm (SM arm) (Other): Patients in this group will receive chemotherapy of gemcitabine and cisplatin only after radiological progression is observed
  Interventions: Drug: gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: gemcitabine — 1,000 mg/m2 intravenous gemcitabine on day 1 and day 8
Drug: Cisplatin — 70 mg/m2 intravenous cisplatin (split into 2 doses on day 1 and day 8)

SUMMARY:
Urothelial carcinomas are one of the most commonly diagnosed cancers worldwide. Postoperative patients carry a poor prognosis with an estimated five-year disease-specific survival rate of 50%. To improve overall survival and reduce the recurrent risk, chemotherapy is recommended as a standard of care. However, currently in Hong Kong, neoadjuvant (preoperational) chemotherapy and adjuvant (postoperative) chemotherapy are not commonly or regularly provided due to the concern of the potential harm from both physicians and patients. Recently, genetic signature from circulating tumor DNA (ctDNA) is emerging as a pivotal biomarker for detecting caner in early stage and molecular residual disease (MRD). With strengths of non-invasive and superior sensitivity, ctDNA is hopefully to serve as a cancer-agnostic surrogate analyte for risk stratification of tumor recurrence, thereby guiding individually tailored treatment. Therefore, this study is proposed to exploratively assess the benefit of ctDNA-guided approach for postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-70 years old;
2. a score of ≤1 for the Eastern Cooperative Oncology Group (ECOG) Performance Status;
3. receiving radical cystectomy (with lymph node dissection) or nephroureterectomy;
4. histologically confirmed (surgical specimen) muscle invasive urothelial carcinoma, and the major histological type should be transitional cell carcinoma;
5. Classification of tumour, node and metastasis (TNM): pT2-4a N0-2M0;
6. absence of microscopic (i.e., positive margin) or gross residual of the tumor (R0 resection) and absence of metastasis, confirmed by a negative CT or MRI scan of pelvis, abdomen and chest within 4 weeks prior to enrolment;
7. adequate hematologic and end-organ function, defined by the following laboratory results obtained within 28 days prior to the first study treatment:

   * ANC≥1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1)
   * WBC counts > 2500 cells/μL
   * Lymphocyte count ≥ 300 cells/μL
   * Platelet count ≥ 100,000 cells/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1)
   * Hemoglobin ≥ 9.0 g/dL
   * AST, ALT, and alkaline phosphatase ≤ 2.5 × the upper limit of normal (ULN),
   * PTT ≤ 1.5 × ULN
   * PT ≤ 1.5 × ULN or INR < 1.7
   * Calculated creatinine clearance ≥ 30 mL/min (Cockcroft-Gault formula)
8. able to understand and provide written informed consent, and agree to receive the treatment arrangement and study procedures stated in the informed consent

Exclusion Criteria:

1. receiving any approved anti-cancer treatment within 3 weeks prior to study enrolment;
2. participation in another clinical trial with therapeutic intent within 28 days prior to enrolment;
3. suffering from malignancies other than urothelial carcinoma within 5 years prior to study enrolment;
4. conditions that contraindicate chemotherapy, such as renal impairment with creatinine clearance rate (CCr) <50 mL/min, hearing impairment, and inadequate marrow function;
5. anaphylactic or hypersensitivity reactions or other contraindication to cisplatin and gemcitabine;
6. active or uncontrolled infections, including human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or tuberculosis;
7. pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the radiational disease-free survival (rDFS) | 1 year

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 1 year
  time to recurrence
Overall Survival (OS) | 5 year
ctDNA clearance rate in ctDNA(+) patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yung Na, PHD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhan Y, Ruan X, Wu Y, Chun TTS, Yao C, Shi R, Liu J, Ali S, Ma R, Huang D, Gao Y, Xu Y, Chen L, Du Q, Ng AT, Li CWB, Xu D, Na R. Surveillance of the Genetic Signature in Circulating Tumor DNA for Guiding Adjuvant Chemotherapy in Urothelial Carcinoma: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 26;14:e72597. doi: 10.2196/72597. PMID 40857715